CLINICAL TRIAL: NCT04480970
Title: Placement of Nasogastric Tubes for Gastric Decompression in Patients With Bronchiolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 261122
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-07

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Nasogastric tube placement (Experimental)
  Interventions: Device: Nasogastric tube placement

INTERVENTIONS:
Device: Nasogastric tube placement — All patients enrolled in the study will have a nasogastric tube placed for gastric decompression.

SUMMARY:
This study aims to evaluate whether placing nasogastric tubes for gastric decompression improves respiratory distress for patients with bronchiolitis who are receiving oxygen via high-flow nasal cannula.

DETAILED DESCRIPTION:
All patients will be consented per IRB procedure. The study will be a prospective study. Study participants will be enrolled after placement on high flow nasal cannula. The respiratory therapist or study staff will use a bronchiolitis scoring tool, the Marlais Risk of Admission Score, to assess the respiratory status of patients after placement on high flow nasal cannula, and prior to placement of NG tube to establish a baseline measurement. This tool includes the following components: respiratory rate, oxygen saturation, heart rate, age, and length of illness. An NG tube will then be placed. Thirty minutes and sixty minutes after placement of the NG tube, the respiratory therapist or study team will again use this scoring tool to assess the respiratory status of the patient. After 60 minutes the study will be concluded. As subject will be requiring oxygen use, admission to an inpatient unit is required. The NG tube will be removed at the discretion of the provider or the admitting physician, who may choose to keep it in at their discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchiolitis by the attending physician
* On high flow nasal cannula (4 liters or greater)
* Ages 0 months to 23 months

Exclusion Criteria:

* Diagnosis of bacterial pneumonia
* History of cranio-facial anomalies
* History of congenital heart disease
* History of G-tube dependence
* History of short gut syndrome
* History of tracheostomy or current tracheostomy

Ages: 1 Day to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory status | 60 minutes
  A bronchiolitis scoring tool, the Marlais Risk of Admission Score, will be used to assess the respiratory status of patients. This tool includes the following components: respiratory rate, oxygen saturation, heart rate, age, and length of illness.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiro, MD, MPH, Principal Investigator — AR Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States